CLINICAL TRIAL: NCT02722291
Title: Functional and Physiological Changes Induced by Pinhole Glasses in Presbyopia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chung-Ang University Hosptial, Chung-Ang University College of Medicine (Other)
Responsible Party: Principal Investigator, Hong Hyun Park, Principal investigator, Chung-Ang University Hosptial, Chung-Ang University College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: ChungAngUHophthalmology
Record Dates: First submitted 2016-03-21; First posted 2016-03-30 (Estimated); Last update posted 2016-04-01 (Estimated); Status verified 2016-03

CONDITIONS: Pinhole
Keywords: presbyopia
MeSH Terms: conditions — Presbyopia

ARMS (1):
- presbyopia (Experimental): All participants perform all exams under 3 conditions, that is baseline, with out pinhole glasses, and with multiple pinhole glasses
  Interventions: Device: Trayner Pinhole Glasses (Trayner Glasses, Ivybridge Devon, U.K.)

INTERVENTIONS:
Device: Trayner Pinhole Glasses (Trayner Glasses, Ivybridge Devon, U.K.)

SUMMARY:
This study is aimed at presbyopic patients that do not require magnifying glass at close rage. The purpose of this study is to investigate the functional and physiological changes in eye induced by pinhole glass.

ELIGIBILITY:
Inclusion Criteria:

1. age over 45 years
2. spherical equivalents(SE) within ± 3.0 diopters(D)
3. normal ocular alignment

Exclusion Criteria:

1. disturbance of accommodation due to any reasons such as an Adie's pupil, Parkinson's disease, a history of previous ocular surgery or trauma, and a history of systemic or topical medication that might affect accommodation
2. corneal pathologic features
3. glaucoma
4. cataracts of grade II or greater by the Lens Opacities Classification System III (LOCS III)
5. vitreous and retinal abnormalities that might limit the accuracy of testing

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-03; Primary Completion 2016-12 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Distant visual acuity (logMAR) | Subjects performed this examination while wearing multiple pinhole and without wearing pinhole with one week apart in random order after baseline study
  Distant visual acuity were measured using Snellen chart (Precision Vision, La Salle, IL, USA) at 4 m.
BUT | Subjects performed this examination while wearing multiple pinhole and without wearing pinhole with one week apart in random order after baseline study
  fluorescein is instilled into the subject's tear film and the subject is asked not to blink while the tear film is observed under a broad beam of cobalt blue illumination
Near point of accommodation (NPA) | Subjects performed this examination while wearing multiple pinhole and without wearing pinhole with one week apart in random order after baseline study
  Near point of accommodation (NPA) was measured using Donder's push-up method.
The fusional convergence | Subjects performed this examination while wearing multiple pinhole and without wearing pinhole with one week apart in random order after baseline study
  With the subject watching the 20/30 sized fixation target at 40 cm, we take the base-out bar prism on the subject's right eye. While gradually increasing the extent of the prism, the first point that the subject noticed diplopia was defined as the break point.
Stereopsis | Subjects performed this examination while wearing multiple pinhole and without wearing pinhole with one week apart in random order after baseline study
  Stereopsis was checked with the Randot Stereotest (Stereo Optical Co., Chicago, IL, USA).
Reading speed (letters per second) | Subjects performed this examination while wearing multiple pinhole and without wearing pinhole with one week apart in random order after baseline study
  Reading speed was evaluated using the famous Korean traditional fairy tale book. This Korean book was printed black-and-white with 10-font size.
Photopic pupil size (baseline, mm) | Subjects performed this examination while wearing multiple pinhole and without wearing pinhole with one week apart in random order after baseline study
  Pupil size under photopic conditions (85 cd/m2) was measured using a WASCA Analyzer (Carl Zeiss Meditec, Oberkochen, Germany).
Pupil size with the one eye pinhole glasses (mm) | Subjects performed this examination while wearing multiple pinhole and without wearing pinhole with one week apart in random order after baseline study
  Pupil size with the one eye pinhole glasses was measured using a WASCA Analyzer (Carl Zeiss Meditec, Oberkochen, Germany).

CONTACTS AND LOCATIONS:
Locations (1):
- Chung-Ang University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Park HH, Park IK, Moon NJ, Chun YS. Clinical feasibility of pinhole glasses in presbyopia. Eur J Ophthalmol. 2019 Mar;29(2):133-140. doi: 10.1177/1120672118810999. Epub 2018 Nov 21. PMID 30460857